CLINICAL TRIAL: NCT03263806
Title: Computed Tomography-derived Fractional Flow Reserve in the Systematic Triage of Emergency Department Acute Chest Pain Patients to Treatment. (The CTFFR-STAT Trial)
Brief Title: The Computed Tomography-derived Fractional Flow Reserve STAT Trial
Acronym: CTFFR-STAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of enrollment
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Gilbert L. Raff, MD, Director Cardiac MRI/CT, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-272
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Heart Disease, Coronary; Chest Pain; Acute Coronary Syndrome
Keywords: angina; coronary artery disease; coronary artery catheterization; coronary CT angiography; fractional flow reserve CT; emergency department
MeSH Terms: conditions — Coronary Disease; Chest Pain; Acute Coronary Syndrome; Angina Pectoris; Coronary Artery Disease; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SOC Group Management (Active Comparator): Attending physicians will dictate SOC management according to their own clinical judgment for medical management, stress test plus imaging or coronary artery catheterization with invasive fractional flow reserve.
  Interventions: Diagnostic Test: SOC Group Management
- CTFFR-Guided Group Management (Experimental): Patients in this group will be triaged using CTFFR. CTFFR values will be provided to physicians with recommendations for medical management or coronary artery catheterization with invasive fractional flow reserve.
  Interventions: Diagnostic Test: CTFFR-Guided Group Management

INTERVENTIONS:
Diagnostic Test: CTFFR-Guided Group Management — Patients will receive standard of care CT on enrollment which will be analyzed by CTFFR. Results will be communicated to the provider who will use CTFFR interpretation to guide care pathway.
  Other Names: Computed tomography - fractional flow reserve
  Arms: CTFFR-Guided Group Management
Diagnostic Test: SOC Group Management — Patients will receive standard of care CT on enrollment which will be analyzed by CTFFR. Results are NOT communicated to the provider who will dictate patient management according to their own clinical judgment
  Arms: SOC Group Management

SUMMARY:
This study is designed to directly compare Standard Care and CT fractional flow reserve (CTFFR) for diagnosis of chest pain patients with definite coronary artery disease (CAD) on heart computed tomography (CT) scans.

DETAILED DESCRIPTION:
New or worsening chest discomfort is the most common symptom of coronary artery disease (CAD), which is plaque build-up in the arteries that supply the heart muscle with blood. Chest pain is one of the most common reasons for emergency department (ED) visits, with an estimated 8 million new cases every year. Evaluation of chest pain is expensive and time consuming, even though 75% of the time it is not due to CAD. It is necessary to carefully define the amount of CAD, even if initial tests reveal no heart attack, because this symptom may progress to heart attack and death if missed.

Coronary artery computed tomography angiography of the heart (CCTA) is one of the most sensitive tests to detect serious CAD in appropriately selected patients.In 85% of acute chest pain (ACP) ED cases tested by CCTA, no CAD or very mild CAD is found, leading to rapid discharge or an alternative diagnosis. However, in the 15% of patients with significant CAD found on CCTA, further evaluation with either stress testing or heart catheterization, and/or hospital admission is required. Since 2015, Beaumont Health hospitals have employed a new FDA-approved test, called CT fractional flow reserve (CTFFR), that can analyze flow down the heart arteries by computer analysis of the original CT images. Results from an analysis of 147 patients suggest that 67% of the time, CTFFR showed no significant flow limitation, providing for the potential to defer invasive testing or treatment for a trial of medical therapy.

The use of CTFFR on ED patients is novel, and it is not yet part of the standard of care (SOC). Standard care of patients with definite CAD on CCTA continues to be hospital admission, stress testing and/or heart catheterization for further diagnosis. Both CTFFR and standard care continue to be used at Beaumont Health, and it is important to determine if one or the other diagnostic strategy is superior. This study is designed to directly compare standard care and CTFFR for diagnosis and management of ACP patients with definite CAD on CCTA.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department chest pain suspicious for ACS based on history and physical examination.
* At least one biomarker (troponin) and electrocardiogram with no evidence of definite ACS.
* A completed CCTA demonstrating >50% but <90% stenosis of at least one coronary artery branch.
* CCTA test images with sufficient diagnostic quality for CTFFR analysis.
* Ability and willingness to provide informed consent.

Exclusion Criteria:

* Left main coronary stenosis of 50% or greater.
* CCTA lesions demonstrating stenosis >90% ("subtotal"), or complex, high-risk plaque characteristics resulting in an a priori recommendation for triage to CATH by the CCTA interpreting physician.
* Attending physician a priori decision for CATH.
* Previous coronary stent, coronary bypass or prior known myocardial infarction.
* Clinical instability, such as hypotension, signs of shock, and/or accelerating chest pain requiring admission.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Raff, MD, Principal Investigator — Beaumont Hospital
Locations (1):
- Beaumont Health System - Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Emergency department patients who had a Cardiac CT scan, were screened for the study. The doctors interpreting the CT scan notifies the research coordinator regarding potential eligibility of the patient to the study.
Period: Overall Study
Arm/Group | SOC Group Management | CTFFR-Guided Group Management
Started | 6 | 7
Completed | 0 (Study Terminated due to lack of enrollment) | 0 (Study Terminated due to lack of enrollment)
Not Completed | 6 | 7
Not completed — Elevated Troponin (failed screen) | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study Termination | 5 | 6

BASELINE CHARACTERISTICS:
Population: Enrolled patients less 1 withdrawal in CTFFR guided group management and 1 patient removed for elevated troponin in SOC group management.
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC Group Management | CTFFR-Guided Group Management | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Median (Full Range); unit: years] | 52 [43 to 76] | 60.5 [47 to 75] | 57 [43 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 4 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Catheterization Rate
Description: Percent of patients undergoing heart catheterization
Time Frame: 3 months after initial presentation
Population: Study terminated with NO data collected.
Arm/Group | SOC Group Management | CTFFR-Guided Group Management
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Diagnostic Effectiveness
Description: Proportion of accurate triage using FFR measured at heart catheterization (CATH-FFR) among all patients triaged to heart catheterization by each strategy
Time Frame: 3 months after initial presentation
Population: Study terminated with NO data collected.
Arm/Group | SOC Group Management | CTFFR-Guided Group Management
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Major Adverse Cardiac Events
Description: Incidence of any serious adverse event, defined as death, acute coronary syndrome or late unscheduled revascularization
Time Frame: 1 year after presentation
Population: Study terminated with NO data collected.
Arm/Group | SOC Group Management | CTFFR-Guided Group Management
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hospital Length of Stay
Description: Time from admission to discharge from hospital in days
Time Frame: An average of 2 days
Population: Study terminated with NO data collected.
Arm/Group | SOC Group Management | CTFFR-Guided Group Management
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | SOC Group Management | CTFFR-Guided Group Management
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

LIMITATIONS AND CAVEATS:
Study terminated early due to difficulty of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT03263806/Prot_SAP_000.pdf